CLINICAL TRIAL: NCT05426369
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Immunogenicity, Preliminary Efficacy and Pharmacokinetics of SCB-219M in the Patients With Chemotherapy-induced Thrombocytopenia
Brief Title: A Clinical Trial Evaluating SCB-219M in in Chemotherapy-induced Thrombocytopenia (CIT)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Clover Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLO-SCB-219M-CHN-001
Record Dates: First submitted 2022-05-10; First posted 2022-06-22 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Chemotherapy-induced Thrombocytopenia (CIT)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose Escalation (Experimental): For single dose escalation, the dose level will be 2µg/kg -15 µg/kg.
  Interventions: Biological: Recombinant Human Tumor Necrosis Factor Receptor II -Fc-TPO Mimetic Peptide Fusion Protein
- Dose Expansion - Group A: First-line CIT treatment / Prophylactic administration for CIT (as needed) (Experimental): The dose level is recommended to be the bioeffective dose obtained from dose escalation and administered once weekly (group A) , with a total of no more than 4 administrations within 70 days after the first dose.
  Interventions: Biological: Recombinant Human Tumor Necrosis Factor Receptor II -Fc-TPO Mimetic Peptide Fusion Protein
- Dose Expansion - Group B: Previously treated or refractory CIT (Experimental): The dose level is recommended to be the bioeffective dose obtained from dose escalation and administered once weekly ( group B ), with a total of no more than 4 administrations within 70 days after the first dose.
  Interventions: Biological: Recombinant Human Tumor Necrosis Factor Receptor II -Fc-TPO Mimetic Peptide Fusion Protein

INTERVENTIONS:
Biological: Recombinant Human Tumor Necrosis Factor Receptor II -Fc-TPO Mimetic Peptide Fusion Protein — Recombinant Human Tumor Necrosis Factor Receptor II -Fc-TPO Mimetic Peptide Fusion Protein for injection (Strength: 1 mg/ml, 0.5ml/vial)

SUMMARY:
A Phase I Clinical Study to Evaluate the Safety, Tolerability, Immunogenicity, Preliminary Efficacy and Pharmacokinetics of SCB-219M in the patients with chemotherapy-induced thrombocytopenia (CIT)

DETAILED DESCRIPTION:
The purpose of this trial is to evaluate the safety, tolerability, immunogenicity, and PK characteristics of single and multiple subcutaneous injections of SCB-219M for CIT, explore the MTD and BED, and preliminarily observe and evaluate efficacy. The trial is divided into a dose escalation phase (Ia) and an expansion phase (Ib).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years (inclusive), voluntary participation with signed informed consent and commitment to protocol-defined visits.
2. Body Weight: ≥40 kg.
3. Diagnosis: Histopathologically/cytopathologically confirmed malignant solid tumors or lymphoma.
4. Phase Ia: Platelet (PLT) & Treatment Status:

<!-- -->

1. PLT <75×10⁹/L during prior chemotherapy cycle;
2. Receiving mono/combination chemotherapy (may include targeted/immunotherapy). 5.Phase Ib: Stratified Requirements:

   * Group A (1st-line CIT prophylaxis/therapy):

<!-- -->

1. PLT <50×10⁹/L, or
2. PLT 50-75×10⁹/L. • Group B (2nd-line CIT therapy/refractory cases): Second-line CIT treatment for refractory or treated CIT patients who failed first-line therapy (rhTPO/IL-11) with platelet count <50×10⁹/L 6.Refractory/Treated CIT Definition:

   * Platelet count remains <50×10⁹/L or increases by <20×10⁹/L within 14 days after completing first-line CIT therapy (e.g., rhTPO or rhIL-11), with baseline PLT <50×10⁹/L at enrollment.

     7.Toxicity Resolution: Prior anti-tumor toxicity ≤ Grade 2 (CTCAE v5.0) at enrollment (alopecia/vitiligo/subjective symptoms excluded).

     8.ECOG PS: 0-2. 9.Life Expectancy: ≥3 months (investigator-assessed). 10.Baseline Laboratory (Pre-dose):
   * a) Creatinine ≤1.5×ULN; CrCl >40 mL/min;
   * b) PT/APTT/INR 80-120% of normal range;
   * c) ANC ≥1.5×10⁹/L;
   * d) Hemoglobin ≥70 g/L;
   * e) Albumin ≥25 g/L. 11.Liver Function:
   * a) ALT/AST ≤3×ULN (≤5×ULN if liver metastasis);
   * b) Total bilirubin ≤2.0×ULN (Gilbert's syndrome/asymptomatic cholelithiasis exempted).

     12.Contraception:
   * Fertile subjects must use ≥1 method:

     o Absolute abstinence;
     * Double-barrier (condom + spermicidal diaphragm);
     * IUD/hormonal contraceptives (oral/implant/patch/injection);
     * Hysterectomy/bilateral salpingectomy/tubal ligation (females or partners);
     * Vasectomy/azoospermia (males or partners).
   * Females: Negative serum β-HCG within 28 days;
   * Males: No sperm donation from first dose to 180 days post-last dose.

Exclusion Criteria:

1. Pregnancy/Lactation: Pregnant or breastfeeding females.
2. Hypersensitivity: Known allergy to protein-based drugs (e.g., recombinant proteins, mAbs) or excipients of the investigational product.
3. Active Infection: Acute infection requiring IV antibiotics without clinical control.
4. Prior Thrombopoietic Agents:

   • Group A: Use within specified windows pre-SCB-219M:

   o Trilaciclib: ≤3 weeks

   o Romiplostim: ≤2 weeks

   o TPO-RAs (e.g., eltrombopag), rhTPO, IL-11, or platelet transfusion: ≤10 days

   • Group B: Use within:

   o Romiplostim/rhTPO/IL-11: ≤7 days

   o TPO-RAs/platelet transfusion: ≤3 days
5. Anticoagulant Use: Anticoagulants/antiplatelet drugs ≤5 half-lives pre-dose or needed during study (aspirin washout ≥7 days).
6. Non-Chemotherapy Thrombocytopenia (within 6 months/unresolved):

1) Clinically significant non-chemotherapy-induced thrombocytopenia (e.g., EDTA-dependent pseudothrombocytopenia) 2) Hematologic malignancies (excluding lymphoma; e.g., leukemia) 3) Multiple myeloma 7.Bleeding Events (within 2 weeks pre-screening):

• Group A: ≥Grade 2 (WHO Bleeding Scale)

* Group B: ≥Grade 3 (WHO Bleeding Scale) 8.Non-CIT Thrombocytopenia Etiologies: 1) Primary immune thrombocytopenia (pITP) 2) Bone marrow failure (e.g., aplastic anemia, Fanconi anemia) 3) Myeloproliferative disorders/MDS 4) Hypersplenism secondary to hematologic/autoimmune diseases 9.Splenectomy/Splenic Effects: Splenic metastasis affecting hematopoiesis; splenectomy/splenic artery embolization ≤12 weeks pre-enrollment.

  10.Uncontrolled Cardiovascular Disease:
* NYHA Class III/IV heart failure
* Pro-thrombotic conditions (e.g., atrial fibrillation, unstable angina)
* QTc >470 ms (>480 ms with bundle branch block)
* Myocardial infarction ≤6 months (Note: Pacemaker/ICD users with normal function eligible) 11.Thrombotic/Coagulation Disorders:
* Coagulopathies
* Arterial/venous thrombosis ≤3 months (excluding PICC-related thrombosis)
* Transient ischemic attack ≤3 months 12.Major Procedures/Radiotherapy: Major surgery/radiotherapy ≤4 weeks pre-dose (except toxicity ≤Grade 2 [CTCAE v5.0], alopecia/vitiligo permitted).

  13.CNS Metastases: Active/untreated CNS or leptomeningeal metastases (asymptomatic brain metastases allowed).

  14.Uncontrolled Hypertension: Resting SBP ≥160 mmHg and/or DBP ≥100 mmHg (two measurements, 2h apart).

  15.Active Infections:
* HIV seropositivity
* Active HBV (HBsAg+ andHBV DNA >LLOQ)
* Active HCV (anti-HCV+ andHCV RNA >LLOQ) 16.Live Vaccines: Live attenuated vaccines ≤4 weeks pre-dose (COVID-19 vaccines permitted except Ad5-vectored type [requires investigator assessment]).

  17.Concurrent Clinical Trials: Participation in other drug/device trials ≤4 weeks pre-dose or planned during study.

  18.Investigator's Discretion: Poor compliance or other factors deemed unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dose escalation: Occurrence of DLT. | Occurrence of DLT from enrollment to day 21.
  Occurrence of DLT
Dose escalation: Frequency of DLT. | Frequency of DLT from enrollment to day 21.
  Frequency of DLT
Dose escalation and Dose expansion:Occurrence of AE. | 28 days after the last administration of SCB-219M
  number, frequency,and charaterization of AEs

SECONDARY OUTCOMES:
Dose escalation: Cmax | up to 21 days after treatment
  Cmax : Maximum serum concentration
Dose escalation: Cmax/D | up to 21 days after treatment
  Cmax/D :Dose normalized Cmax
Dose escalation: tmax | up to 21 days after treatment
  tmax : Time to Cmax
Dose escalation: AUC0-24h | up to 21 days after treatment
  AUC0-24h: Area under the serum concentration-time curve from 0 h to 24 h
Dose escalation: AUC0-last | up to 21 days after treatment
  AUC0-last :Area under the serum concentration-time curve from 0 h on Day 1 to the last time point with a quantifiable concentration
Dose escalation: AUC0-inf | up to 21 days after treatment
  AUC0-inf : Area under the serum concentration-time curve from 0 h extrapolated to infinity
Dose escalation: t1/2 | up to 21 days after treatment
  t1/2 : Apparent half-life
Dose escalation: CL/F | up to 21 days after treatment
  CL/F: Systemic clearance
Dose escalation: Vz/F | up to 21 days after treatment
  Vz/F: Volume of distribution
Dose escalation: λz | up to 21 days after treatment
  λz: Elimination rate constant
Dose escalation: Preliminary efficacy assessment.The percentage of subjects requiring platelet infusion and the frequency of infusion during the DLT observation period. | up to 28 days after administration
  The percentage of subjects requiring platelet infusion and the frequency of infusion during the DLT observation period.
Dose escalation: Preliminary efficacy assessment. | up to 28 days after administration
  Duration of PLT count ≥50×10^9/L and percentage of subjects during the DLT observation period.
Dose escalation: Preliminary efficacy assessment. | up to 28 days after administration
  Duration of PLT count ≥75×10^9/L and percentage of subjects during the DLT observation period.
Dose escalation: Preliminary efficacy assessment. | up to 28 days after administration
  Duration of PLT count ≥100×10^9/L and percentage of subjects during the DLT observation period
Dose expansion:：PK parameters of SCB-219M were established after repeated abdominal subcutaneous injections. | up to 168 hours after the last treatment
  The PK parameters include: C₀, Cmax/D, Css_min, Cmax_ss, Cav_ss, Rac, tmax, AUC₀-last, AUC₀-inf, AUCss, DF, MRT, t₁/₂, etc.
Dose expansion: Preliminary efficacy assessment. | 28 days after the last administration of SCB-219M
  Incidence of grade 2/3/4 thrombocytopenia (CTCAE version 5.0).
Dose expansion: Preliminary efficacy assessment. | Within 7, 14, 21, and 28 calendar days post-administration
  Percentage of subjects requiring platelet transfusions and number of transfusions within 7, 14, 21, and 28 days post-dose
Dose expansion: ：Platelet response onset time (days), duration of platelet effect maintenance (days), and overall response rate (%). | 28 days after the last administration of SCB-219M
  Key efficacy endpoints per protocol:
  1. Time (days) to first achievement of platelet counts ≥50×10⁹/L, ≥75×10⁹/L, and ≥100×10⁹/L post-dose ;;
  2. Duration (days) of sustained platelet count maintenance at or above prespecified thresholds (≥50×10⁹/L, ≥75×10⁹/L, ≥100×10⁹/L);
  3. Responder rate (%) , defined as the proportion of subjects achieving predefined platelet count thresholds.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China